CLINICAL TRIAL: NCT06895356
Title: A Phase 1, Two Part, Randomized, Single and Multiple Dose Crossover Study to Assess the Relative Bioavailability Between Tavapadon Clinical and Commercial Tablets
Brief Title: A Study to Assess the Relative Bioavailability of Oral Tavapadon in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M25-974
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tavapadon: Part 1-Sequence 1 (Experimental): Participants will receive Clinical Tavapadon Dose A in Period 1, followed by Commercial Tavapadon Dose B in Period 2
  Interventions: Drug: Tavapadon
- Tavapadon: Part 1-Sequence 2 (Experimental): Participants will receive Commercial Clinical Tavapadon Dose B in Period 1, followed by Clinical Tavapadon Dose A in Period 2
  Interventions: Drug: Tavapadon
- Tavapadon: Part 2-Sequence 1 (Experimental): Participants will receive Clinical Tavapadon Dose C in Period 1, Clinical Tavapadon Dose D in Period 2 followed by Commercial Tavapadon Dose E in Period 3
  Interventions: Drug: Tavapadon
- Tavapadon: Part 2-Sequence 2 (Experimental): Participants will receive Clinical Tavapadon Dose C in Period 1, Commercial Tavapadon Dose E in Period 2 followed by Clinical Tavapadon Dose D in Period 3
  Interventions: Drug: Tavapadon

INTERVENTIONS:
Drug: Tavapadon — Oral: Tablet

SUMMARY:
This study will assess the relative bioavailability of two different Oral formulations of tavapadon in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal at the time of screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG
* Females, Non-Childbearing Potential due to meeting the following criteria:

  * Permanent sterility due to a hysterectomy, bilateral salpingectomy, bilateral oophorectomy.
  * Non-surgical permanent infertility due to Mullerian agenesis, androgen insensitivity, or gonadal dysgenesis; investigator discretion should be applied to determining study entry.
  * Postmenopausal female who is age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND a follicle-stimulating hormone (FSH) level ≥ 30 IU/L.

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of suicidal ideation within one year prior to study drug administration as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity rating scale (C-SSRS) completed at Screening, or any history of suicide attempts within the last two years.
* Use of tobacco- or nicotine-containing products within 90 days prior to the first dose of study treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 53 days
  An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment
Maximum Observed Plasma Concentration (Cmax) of Tavapadon | Up to approximately 22 days
  (Cmax) of Tavapadon
Time to Cmax (Tmax) of Tavapadon | Up to approximately 22 days
  Tmax of Tavapadon
Apparent Terminal Phase Elimination Rate Constant (β) of Tavapadon | Up to approximately 22 days
  Apparent Terminal Phase Elimination Rate Constant (β) of Tavapadon
Terminal Phase Elimination Half-life (t1/2) of Tavapadon | Up to approximately 22 days
  Terminal Phase Elimination Half-life (t1/2) of Tavapadon
Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUCτ) of Tavapadon | Up to approximately 22 days
  Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUCτ) of Tavapadon
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Tavapadon | Up to approximately 22 days
  Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Tavapadon
Trough Concentration (Ctrough) of Tavapadon | Up to approximately 22 days
  Trough Concentration (Ctrough) of Tavapadon

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 275870, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-974